CLINICAL TRIAL: NCT02996435
Title: smartADHERE - Smartphones to Improve Rivaroxaban ADHEREnce in Atrial Fibrillation
Brief Title: Smartphones to Improve Rivaroxaban ADHEREnce in Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108260; 39039039AFL4010 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Adherence Platform (Experimental): Participant adherence will be monitored using a mobile application and platform which provides a real-time reminder that alerts the participant to take his or her medication. The application will also send an alert to the participant when a refill is needed based on calculated medication or pill supply. The intervention will focus only on daily adherence to rivaroxaban.
  Interventions: Behavioral: Mobile Application Intervention
- Control: Standard of Care (Other): Participants will receive physician- or nurse-guided standard of care for their rivaroxaban adherence. No drug will be administered as part of this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Behavioral: Mobile Application Intervention — Mobile phone application that sends reminders and allows participants to self-manage their medication adherence. Monitoring of participant adherence from this tool will be performed by the central coordinating center, which will send notifications or contact the participant based on the adherence history in accordance with the study protocol.
  Other Names: Care4Today®
  Arms: Mobile Adherence Platform
Other: No Intervention — Participants will receive physician- or nurse-guided standard of care.
  Arms: Control: Standard of Care

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness of an intervention with a mobile adherence platform, compared to physician- or nurse-guided standard of care, to improve medication adherence to rivaroxaban in participants who have recently initiated treatment with rivaroxaban for stroke prevention in atrial fibrillation based on an assessment of the proportion of days covered (PDC) of rivaroxaban treatment.

ELIGIBILITY:
Inclusion Criteria:

* A history of atrial fibrillation
* Taking newly-prescribed rivaroxaban for atrial fibrillation for less than or equal to (<=) 90 days or who are about to initiate therapy (with a prescription dated in the last 90 days)
* At least 1 of the 4 questions answered "yes" from the four-item Morisky Medication Adherence Scale (MMAS-4)
* Possession of a compatible smartphone with an active phone number, text and data plan. The smartphone must be in continued possession of the participant. It may not be a shared device and must exclusively remain in the possession of the participant during the study period. The smartphone must have an active cellular phone number and cellular data subscription. WiFi internet capability is not a substitute for an active cellular data plan
* Willing to have the adherence application installed on a smartphone and use it every day during the entire study period
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study and is willing to authorize the study team to contact the participant's pharmacy for oral anticoagulation medication and refill data
* Willing to provide oral confirmation indicating that he/she has not previously used a medication adherence application
* Ability to read and understand English

Exclusion Criteria:

* Anticipated inability to adhere to the mobile application (Care4Today) based on opinion of site Principal Investigator (PI)
* Anticipated rivaroxaban use less than (<) 12 months based on clinical documentation or participant interview
* Prescribed rivaroxaban for indications other than atrial fibrillation (Prescriptions for concomitant conditions are allowed as long as 1 of the indications is atrial fibrillation)
* Current use of: specialized anticoagulation clinics for rivaroxaban medication management; specialized pharmacist-led adherence or refill monitoring; or enrollment in a medication adherence program even if that program is for medications other than rivaroxaban
* Current use of adherence tracking devices, hardware, smartphone or computer applications, including but not limited to smart pill bottles, pill timers, radiofrequency tagged medications or dispensers, mobile applications, or automated phone reminders. Pharmacy and health care plan automated refill reminders are permitted and are not exclusion. Pill organizers or containers that only compartmentalize a participant's medications based on days of the week are not exclusion. Pill organizers that remind participants when to take medicine with beeps or alerts are exclusion
* Cognitive, visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of mobile phone
* Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Proportion of Days Covered (PDC) | Month 6
  Adherence to rivaroxaban medication will be estimated based on validated PDC algorithm. PDC (expressed as percentage) defined as non-hospitalized days during which oral anticoagulant (OAC) will be supplied and consumed over total observation time duration during which rivaroxaban should have been consumed.

SECONDARY OUTCOMES:
Percentage of Participants With PDC Greater Than or Equal to (>=) 80 Percent | Month 6
  PDC defined as non-hospitalized days during which oral anticoagulant (OAC) will be supplied and consumed over total observation time duration during which rivaroxaban should have been consumed.
Change From Baseline in the Average Score on the Eight-item Morisky Medication Adherence Scale (MMAS-8) | Month 6
  The MMAS-8 scale is a recognized indicator of medication adherence, consisting of 8 questions with a sum score ranging between 0 and 8 points. The higher score indicates higher adherence to the prescribed therapy recommendation.
Measure of Medication Persistence of Rivaroxaban | Month 6
  Measure of medication persistence of rivaroxaban defined as the percentage of participants on rivaroxaban with an active prescription at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (25):
- United States (25):
  - Anchorage, Alaska
  - Los Angeles, California
  - Manhattan Beach, California
  - Oakland, California
  - Pasadena, California
  - Stanford, California
  - Ventura, California
  - Pensacola, Florida
  - Overland Park, Kansas
  - Lexington, Kentucky
  - Saint Joseph, Michigan
  - Reno, Nevada
  - Buffalo, New York
  - Jamaica, New York
  - Lake Success, New York
  - Mineola, New York
  - Saratoga Springs, New York
  - Canton, Ohio
  - Doylestown, Pennsylvania
  - Reading, Pennsylvania
  - Yardley, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Bellevue, Washington

REFERENCES:
- [Derived] Turakhia M, Sundaram V, Smith SN, Ding V, Michael Ho P, Kowey PR, Piccini JP, Foody J, Birmingham MC, Ianus J, Rajmane A, Mahaffey KW; smartADHERE Investigators. Efficacy of a centralized, blended electronic, and human intervention to improve direct oral anticoagulant adherence: Smartphones to improve rivaroxaban ADHEREnce in atrial fibrillation (SmartADHERE) a randomized clinical trial. Am Heart J. 2021 Jul;237:68-78. doi: 10.1016/j.ahj.2021.02.023. Epub 2021 Mar 4. PMID 33676886